CLINICAL TRIAL: NCT04301102
Title: Intraoperative Hemodynamic Optimization Using the Hypotension Prediction Index and Its Impact of Tissular Perfusion
Brief Title: The Predict H Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Juan Victor Lorente (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor-Investigator, Juan Victor Lorente, Anesthesiologist, Andalusian Network for Design and Translation of Advanced Therapies
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: v 1.0; March 2019
Record Dates: First submitted 2020-02-19; First posted 2020-03-10 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Intraoperative Hypotension
Keywords: goal directed hemodynamic therapy; machine learning; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Hemodynamic management will be based on the functional hemodynamic parameters provided by Hemosphere platform with the Acumen IQ sensor, including cardiac output, stroke volume, SVV and Acumen IQ specific parameters: maximal arterial pressure rise (dP/dtmax), dynamic arterial elastance (Eadyn) and HPI
  As a pattern replacement of interstitial space, we will use balanced crystalloid (Isofundin®) at 1-3 ml / kg / h in case of laparoscopic surgery and 5 to 7 ml / kg / h in case of open surgery.
  The protocol of action on the intravascular space will be based on the maintenance of systolic volume with colloids (hydroxyethyl starch - Voluvén®).
  Interventions: Device: Hemosphere platform® together with the FloTrac Acumen IQ® sensor
- Control (Other): Hemodynamic management will be based on the functional hemodynamic parameters provided by the HemoSphere platform® with the FloTrac® sensor, including cardiac output (CO), stroke volume (SV), and stroke volume variation (SVV)
  As a pattern replacement of interstitial space, we use balanced crystalloid (Isofundin®) at 1-3 ml / kg / h in case of laparoscopic surgery and 5 to 7 ml / kg / h in case of open surgery.
  The protocol action for the intravascular space will be based on a recently published hemodynamic optimization algorithm (Heming N, Moine P, Coscas R, Annane D. Perioperative fluid management for major elective surgery. British Journal of Surgery. 2020;107:e56-62). The fluid used will be hydroxyethyl starch (Voluven®).
  Interventions: Device: Hemosphere platform® together with the FloTrac® sensor

INTERVENTIONS:
Device: Hemosphere platform® together with the FloTrac Acumen IQ® sensor — Clinical platform that, analyzing the pulse wave contour, obtained from the previously catheterized radial artery, is able to make available to the clinician both a continuous monitoring of blood pressure and advanced hemodynamic parameters that help patient management. It incorporates predictive parameters such as the hypotension prediction index and decision support parameters such as dynamic arterial elastance and maximum dP / dT.
  It also has the possibility of assessing regional oxygen saturation, measured by near-infrared light photoplethysmography, and the sensor can be applied in different locations (cerebral, muscular ...).
  Arms: Experimental
Device: Hemosphere platform® together with the FloTrac® sensor — Clinical platform that, analyzing the pulse wave contour, obtained from the previously catheterized radial artery, is able to make available to the clinician both a continuous monitoring of blood pressure and advanced hemodynamic parameters that help patient management.
  It also has the possibility of assessing regional oxygen saturation, measured by near-infrared light photoplethysmography, and the sensor can be applied in different locations (cerebral, muscular ...).
  Arms: Control

SUMMARY:
The aim of the study is to determine whether a goal-directed algorithm based on the prevention of arterial hypotension using the Hypotension Prediction Index reduces the duration and severity of intraoperative hypotension when compared with the recommended standard therapy and if this intraoperative strategy affects tissue oxygenation and organ perfusion.

DETAILED DESCRIPTION:
Background: Intraoperative arterial hypotension is associated with poor postoperative outcomes. The Hypotension Prediction Index developed from machine learning, predicts the occurrence of arterial hypotension from the analysis of the arterial pressure waveform. The use of this index can reduce the duration and severity of intraoperative hypotension in adults undergoing noncardiac surgery.

Methods: We will conduct a multicenter, randomized, controlled trial (N=80) in high-risk surgical patients scheduled for elective major abdominal surgery. All participants will be randomly assigned to a control or intervention group. Hemodynamic management in the control group will be based on standard hemodynamic parameters. Hemodynamic management of patients in the intervention group will be based on functional hemodynamic parameters provided by Hemosphere platform (Edwards Lifesciences Ltd), including dynamic arterial elastance, dP/dtmax and the Hypotension Prediction Index. Tissue oxygen saturation will be non-invasively and continuously recorded by using near-infrared spectroscopy technology. Biomarkers of acute kidney stress (cTIMP2 and IGFBP7) will be obtained before and after surgery. The primary outcome will be intraoperative time-weighted average with a mean arterial pressure < 65mmHg.

Discussion: The aim of the study is to determine whether a goal-directed algorithm based on the prevention of arterial hypotension using the Hypotension Prediction Index reduces the duration and severity of intraoperative hypotension when compared with the recommended standard therapy and if this intraoperative strategy affects tissue oxygenation and organ perfusion.

ELIGIBILITY:
Enrolled patients will be at least 65 years old and/or American Society of Anesthesiologist (ASA) physical status III/IV, scheduled for elective major abdominal surgery (general surgery, urology, or gynecology, through laparoscopic or open approach), with general or combined anesthesia. Surgery will be considered to be major if the expected duration is > 2 h, or the estimated blood loss is > 15% of blood volume, or if the expected required transfusion is ≥ 2 packed red blood cells.

Exclusion criteria will be pregnancy, surgery performed only under regional anesthesia, preoperative glomerular filtrate < 60 ml/min/1.73m2 according to the CKD-EPI 2009 formula, persistent atrial fibrillation, known cardiac shunts or if the patient received a kidney transplant, and refusal of the patient to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
TWA-MAP< 65 mmHg | Intraoperatively
  Area between 65 mmHg threshold and the curve of the MAP measurements divided by the total continuous reading time mmHg for a minimum duration of 1 minute (3 consecutive records from one minute to more between two consecutive falls).
Number of intraoperative hypotension episodes | Intraoperatively
  defined as an event of MAP < 65 mmHg of at least 1-minute duration
Total time of hypotension per case | Intraoperatively
  Intraoperative Total time of hypotension (MAP < 65 mmHg)

SECONDARY OUTCOMES:
StO2 | Intraoperatively
  StO2 will be non-invasively and continuously recorded in the brachioradial muscle in the arm opposite to the arterial line. We calculated the time averaged StO2 per patient and identified the minimum StO2, defined as the minimum value sustained (+1%) over at least 5 min
Acute kidney stress biomarkers | NC1: after anestesic induction // NC2: First 4 hours after the patient is admitted to the UCI/REA // NC3: 12 hours after NC2.
  Urine immunoassay, commercially known as Nephrocheck® (Biomerieux). The first sample (NC1) will be collected after anesthetic induction, when performing bladder catheterization. The first postoperative sample (NC2) will be collected during the first 4 hours after the patient is admitted to the UCI / REA for their postoperative stay. If the AKIRisk value in that first postoperative sample (NC2) is less than 0.3, no new Nephrocheck® determinations will be collected. If the AKIRisk value in the first postoperative sample (NC2) is greater than 2, no further Nephrocheck® determinations will be made. If the AKIRisk value in that first postoperative sample (NC2) is between 0.3 and 2, we will collect a second postoperative sample (NC3) at 12 hours of the first. No more Nephrocheck® determinations will be made.
Postoperative complications | Postoperatively
  The analysis of postoperative complications will be carried out in accordance with European EPCO recommendations.
Length of hospital stay | At 30 days
Mortality | At 30 days
Total fluid therapy during surgery | Intraoperatively
  Types and total amounts
Accumulated dose of Fentanyl, remifentanyl and/or morphine. | Intraoperatively
  Accumulated dose during the intraoperative period
Accumulated dose during the intraoperative period of vasoactive | Intraoperatively
  Specify by drugs used and method of infusion (bolus / continuous infusion pump)
Accumulated dose during the intraoperative period of ionotopic drug | Intraoperatively
  In case of indication.
Need and accumulated dose of drugs not included in previous groups | Intraoperatively
  Dexmedetomidine, esmolol or other drugs with hemodynamic impact
Transfusion of total blood products during surgery | Intraoperatively

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitario Juan Ramón Jiménez, Huelva
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in sickle cell anemia. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact juanvictor.lorente@gmail.com

REFERENCES:
- [Derived] Lorente JV, Jimenez I, Ripolles-Melchor J, Becerra A, Wesselink W, Reguant F, Mojarro I, Fuentes MLA, Abad-Motos A, Agudelo E, Herrero-Machancoses F, Callejo P, Bosch J, Monge MI. Intraoperative haemodynamic optimisation using the Hypotension Prediction Index and its impact on tissular perfusion: a protocol for a randomised controlled trial. BMJ Open. 2022 Jun 2;12(6):e051728. doi: 10.1136/bmjopen-2021-051728. PMID 35654467